CLINICAL TRIAL: NCT04298242
Title: A Phase I Study of Magnetic Resonance Guided High Intensity Focused Ultrasound for Treatment of Advanced Pancreatic Adenocarcinoma
Brief Title: Magnetic Resonance Guided High Intensity Focused Ultrasound in Advanced Pancreatic Adenocarcinoma Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-52567; PANC0034 (Other: OnCore); NCI-2020-13809 (Other: CTRP)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRgFUS Treatment (Experimental): The pancreatic tumor will be ablated with magnetic resonance guided focused ultrasound (MRgFUS).
  Interventions: Device: ExAblate 2100

INTERVENTIONS:
Device: ExAblate 2100 — A non-invasive thermal ablation device fully integrated with an MR imaging system
  Other Names: InSightec ExAblate 2100 MRgHIFU system

SUMMARY:
The primary purpose of this protocol is to assess the ExAblate 2100 MR guided high intensity focused ultrasound device as an intervention for treatment of advanced stage pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Primary Objective: The primary endpoints for this study will be 1) feasibility of ablation and 2) safety of ablation.

Secondary Objective: 1.)Pain reduction after ablation. 2.) Evidence of inflammation at ablation site based on histology, or in blood after ablation

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Patients willing to sign a written informed consent document
* Patients with unresectable, locally advanced or metastatic pancreatic adenocarcinoma
* Patients with upper abdominal pain rating at least 4 out of 10 in severity on BPI
* Tumor must be visualized on CT or MRI, obtained within 30 days of enrollment
* Tumor must be accessible to the ExAblate MRgFUS device
* Life expectancy ≥ 3 months, as determined by oncologist and documented in chart
* ECOG performance status of 0, 1, or 2
* INR < 1.6, platelet count > 50,000 microL
* Serum urate, calcium, potassium, phosphate, creatinine < 1.5x upper limit of normal
* Patients can receive general anesthesia, as determined by anesthesiologist

Exclusion Criteria:

* Previous pancreatic surgery
* Patients with contraindication for MR imaging such as implanted metallic devices that are not MRI-safe, size limitations, claustrophobia, etc.
* Patients with known intolerance or allergy to MR contrast agent (gadolinium chelates) including advanced kidney disease (GFR <30 mL/min/1.73 m2) or on dialysis
* Pregnant and nursing patients will be excluded from the study because of a contraindication to administering MRI contrast agents to these patients
* Patients unable to receive general anesthesia
* Target is:

  1. NOT visible by non-contrast MRI, OR
  2. NOT accessible to ExAblate device
* Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (can be up to 6 hrs of total table time)
* Patients with acute medical condition (e.g. pneumonia, sepsis) that is expected to hinder them from completing this study
* Patients with unstable cardiac status including:

  1. Unstable angina pectoris on medication
  2. Patients with documented myocardial infarction within six months of protocol entry
  3. Congestive heart failure requiring medication (other than diuretic)
  4. Patients on anti-arrhythmic drugs
  5. Patients with severe hypertension (diastolic BP > 100 on medication)
  6. Patients with severe hematologic, neurologic, or other uncontrolled disease (e.g. platelets < 50,000/microL, INR > 1.5)
* Patients who are taking anti-thrombotic medication
* Severe cerebrovascular disease (multiple CVAs or CVA within 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Measure acceptable ablation percentage | Immediately after MRgFUS treatment
  Feasibility of ablation, as measured by the number of patients with acceptable ablation percentage. Acceptable ablation percentage is defined as ≥50% of the targeted volume appearing ablated on post-treatment imaging. Ablation will be deemed feasible if at least seven of the ten patients have an acceptable ablation percentage
Total frequency and severity of adverse events | 24 months
  Safety of ablation, as measured by the total frequency and severity of adverse events. Adverse events will be categorized and grade for severity according to the Common Terminology Criteria for Adverse Events, Version 5.0. Ablation will be deemed safe if there are no treatment-related serious adverse events, and no more than five moderate or mild treatment-related adverse events, among the ten patients during follow up.

SECONDARY OUTCOMES:
Assess Pain Response assessed by the Brief Pain Inventory (BPI) | Baseline, 1 week, and monthly for 24 months following treatment
  Reduction in pain level, as measured by:
  a. a decline in pain score after one week of at least 2 points, or a pain score < 4 out of 10, as assessed by the Brief Pain Inventory. Ablation will be deemed pain reducing if at least five of the ten patients have pain reduction.
Assess Pain Response assessed by morphine equivalent daily dose (MEDD) | Baseline, 1 week, and monthly for 24 months following treatment
  Reduction in pain level will be measured by a decline after one week in morphine equivalent daily dose (MEDD) of 25%. Ablation will be deemed pain reducing if at least five of the ten patients have pain reduction.
Evidence of ablation-induced inflammation | 1week
  Evidence of ablation-induced inflammation, defined as post-ablation increases in histologic and/or blood measures of inflammation markers, as measured by either:
  1. an increase in tumor infiltrating CD8+ T cells
  2. a decrease in immune suppressive cells (Tregs, macrophages) in the tumor
  3. an increase in immune activation signatures (including interferon gamma) in the tumor as measured by RNAseq
  4. a change in immune profile in the circulating immune cells (PBMCs) to reflect an activated immune response (e.g. activated T or B cells, reduction in immune suppressive cells or cytokines) Ablation will be deemed inflammation-inducing if at least five of the ten patients show at least a 50% increase in inflammation on at least 2 of the 4 markers

CONTACTS AND LOCATIONS:
Overall Officials: Pejman Ghanouni, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No